CLINICAL TRIAL: NCT05644067
Title: A Randomised, Controlled, Double-blind, Parallel Group, Single Center Phase Ib Trial to Assess Safety, Reactogenicity and Immunogenicity of a Candidate Dual-stage Malaria Vaccine, SumayaVac-1 (MSP-1 With GLA-SE as Adjuvant) in Healthy Malaria Exposed Adults of African Origin Aged 18-45 Years
Brief Title: Assessment of the Malaria Vaccine Candidate SumayaVac-1 in Healthy Adults Aged 18-45 Years Living in a Malaria Endemic Country
Acronym: SUM-101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Ifakara Health Institute (Other); Sumaya Biotech GmbH & Co. KG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: P2267-22
Record Dates: First submitted 2022-10-27; First posted 2022-12-09 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2022-10

CONDITIONS: Malaria
Keywords: Plasmodium falciparum; MSP-1; Tanzania; Phase Ib; Vaccine; GLA-SE
MeSH Terms: conditions — Malaria; Malaria, Falciparum

STUDY DESIGN:
Intervention Model Description: A randomised, controlled, double-blind, parallel group, single center Phase Ib trial to assess safety, reactogenicity, immunogenicity of a candidate dual-stage malaria vaccine, SumayaVac-1 (MSP-1 with GLA-SE as adjuvant) in healthy participants aged 18-45 years.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial will be conducted in a double-blinded manner. Namely, the participants, site staff, sponsor staff, the study monitor(s) and the trial statistician will be blinded to the treatment allocation. The independent statistician and the pharmacist are not blind throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SumayaVac-1(SUM-101) (Experimental): Candidate malaria Vaccine (Investigational Medicinal Product (IMP)). 20 participants will be randomised to receive three monthly inoculations of the IMP
  Interventions: Biological: SumayaVac-1(SUM-101)
- Verorab (Placebo Comparator): Comparator used as a control. 20 participants will be randomised to receive three monthly inoculations of the comparator.
  Interventions: Biological: Verorab

INTERVENTIONS:
Biological: SumayaVac-1(SUM-101) — One immunization every 4 weeks for 3 months (total 3 immunizations)
  Arms: SumayaVac-1(SUM-101)
Biological: Verorab — One immunization every 4 weeks for 3 months (total 3 immunizations)
  Arms: Verorab

SUMMARY:
Malaria remains a major infectious disease causing a heavy burden of mortality and morbidity in populations living in tropical and subtropical regions. Large, international research efforts have been invested into the development of anti-malaria vaccination strategies, however, currently there is only one malaria vaccine approved for use in the pediatric population, which provides a moderate and short-lived protection. Therefore, there is a need to develop a malaria vaccine that will be essential to further strengthen malaria control measures in future.

A Phase Ia trial with the same IMP (SumayaVac-1 vaccine developed using a full-length recombinant MSP-1 administered along with the adjuvant GLA-SE) in Caucasians in Heidelberg, Germany, proved to be well tolerated and safe. However, a Phase Ib clinical trial on healthy participants residing in a malaria endemic country would be essential to evaluate the safety and reactogenicity in the target population. The project aims to investigate the safety, reactogenicity, immunogenicity of the candidate malaria vaccine, SumayaVac-1 (SUM-101) in 40 healthy participants (men and women) of African origin in Bagamoyo, Tanzania.

DETAILED DESCRIPTION:
Objectives:

To evaluate in healthy adults of African origin previously exposed to the malaria parasite receiving SumayaVac-1 (SUM-101) versus rabies control (Verorab®) vaccine:

Primary Objectives

* Safety and reactogenicity of SumayaVac-1 (SUM-101).
* Immunogenicity of SumayaVac-1 (SUM-101).

Secondary Objectives

• SumayaVac-1 (SUM-101) vaccine-induced antibody levels, in vitro effector functions.

Exploratory Objectives

* Comparison of SumayaVac-1 (SUM-101) induced immunoglobulin isotype distribution and duration between malaria pre-exposed and malaria naïve participants from the previous Phase Ia study in Heidelberg.
* Fine scale epitope mapping of SumayaVac-1 (SUM-101) specific antibodies using peptide arrays, to investigate humoral immune response at baseline with vaccine induced responses.
* Comparison of SumayaVac-1 (SUM-101) induced cellular immunity between malaria pre-exposed and malaria naïve participants from the previous Phase Ia study in Heidelberg including fine scale epitope mapping of MSP-1 specific CD4+ and CD8+ T cells.
* Investigation of the B- and T-Cell repertoire before and after SumayaVac-1 (SUM-101) vaccination.
* Integrated transcriptome and immunoglobulin gene repertoire analyses of MSP-1 specific B-cells using single-cell technologies.
* Glycosylation patterns of MSP-1 specific functional antibodies.
* Investigate off-target IgG and IgM repertoire after SumayaVac-1 (SUM-101) vaccination using immunoproteomics.
* Investigate the structure of MSP-1 protein bound to functional antibodies by cryo-electron tomography to map conformational epitopes.
* To evaluate mechanisms of malaria specific antibody diversity generation, post-translational modification of antibodies, and B- and T-cell memory generation and maintenance.
* Ex vivo assessment of changes in human peripheral blood transcriptome in participants having received SumayaVac-1 (SUM-101) versus Verorab® rabies vaccine.
* Description of ɣδ T-cell receptor repertoire, transcriptome, functional activity and phenotypes in participants having received SumayaVac-1 (SUM-101) versus Verorab® rabies vaccine.
* Investigate impact of presence of intestinal helminth infections on SumayaVac-1(SUM-101) induced humoral immune response.
* Investigate impact of presence of intestinal helminth infections on SumayaVac-1(SUM-101) induced cellular immune response.

Study Design:

This is a randomised, controlled, double-blind, parallel group, single center Phase Ib trial to assess the safety, reactogenicity, and immunogenicity of SumayaVac-1 (SUM-101) in healthy, malaria-exposed adults of African origin aged 18-45 years.

In total, 40 participants will be enrolled (male and female). 20 participants will be randomised to receive three monthly inoculations (on D0, D28 and D56) with the investigational product, SumayaVac-1 (SUM-101), and 20 participants will be randomised to receive the registered rabies vaccine, Verorab®, as controls.

For operational reasons the participants will be split in two groups of 20 participants.

* Group 1 will have a sentinel subgroup (2 SumayaVac-1 (SUM-101) & 1 Verorab® rabies vaccine) with a 48 hours safety surveillance period before the remaining 17 participants (8 SumayaVac-1 (SUM-101) & 9 Verorab® rabies vaccine) of the group 1 receive their 1st vaccination.
* Group 2 will be composed of 20 participants (10 SumayaVac-1 (SUM-101) & 10 Verorab® rabies vaccine). All visits in group 2 will be shifted by at least 3 weeks compared to group 1 to create minimal overlap of study-related activities.

After each vaccination (done on D0, D28 and D56), the participants will remain at the facility for 2 hours prior to their discharge for home. The participant will be called daily by phone (or home visits if required) until 6 days post vaccination for follow-up.

For all participants, vaccination follow-up visits at the site will occur at 7, 14 and 28 days after each vaccination.

Measurements and Procedures:

Written informed consent will be taken prior to any study procedure. Healthy participants will be screened and randomised before administration of the study IMP.

On the day of the 1st vaccination, the health status of the participant is re-checked and eligibility confirmed. Samples for safety, humoral, cellular and exploratory measurements are taken before 1st vaccination (baseline). Vaccination is administered and the participant remains at site for 2 hours before being discharged. Telephone follow-ups (or home visits if required) will be performed daily until 6 days after each vaccination. On 7, 14 and 28 days after each vaccination (done on D0, D28 and D56), the participant will be invited to come back to the facility and health status is checked.

Further participant follow-up visits will take place at D112 (W16) and D140 (W20) post 1st vaccination. Sampling for humoral and cellular responses will be performed at D112 (W16) and D140 (W20). Additionally, sampling for exploratory measurements will be performed at D112 (W16) (Vac1 + 4 month follow-up site visit).

Number of Participants with Rationale:

Vaccination: 40 adult participants Overall: 20 SumayaVac-1 (SUM-101) and 20 Verorab® control

Group 1 Sentinel sub-group

* 2 SumayaVac-1 (SUM-101)
* 1 Verorab® control

Group 1 Follower Group

* 8 SumayaVac-1 (SUM-101)
* 9 Verorab® control

Group 2

* 10 SumayaVac-1 (SUM-101)
* 10 Verorab® control

As this is a Phase I trial, no formal sample size calculation has been done. The sample size is considered sufficient to examine the safety and reactogenicity of SumayaVac-1 (SUM-101), and humoral and cellular immunogenicity.

Study Product / Intervention:

Vaccination: Intra-muscular injection of SumayaVac-1 (SUM-101) composed of 150 µg MSP-1 drug product + 5 μg GLA-SE adjuvant CHMI: Direct venous inoculation of 3.2 x 103 purified, infectious P. falciparum sporozoites

Control Intervention: Vaccination control: Intra-muscular injection of rabies vaccine (Verorab®)

Study Duration: The total study duration including the screening period (~4 weeks) combining Group 1 and 2 will be approximately 35 weeks.

The study duration for each participant will be ~24 weeks (4 weeks of screening period plus 20 weeks of vaccinations and long-term follow-up visits).

Study Centre: The Ifakara Health Institute Bagamoyo Clinical Trial Facility.

Statistical Analysis incl. Power Analysis:

See above for sample size justification. To evaluate the safety and reactogenicity primary endpoints, AEs and SAEs will be presented according to the endpoint definitions above. AE reporting will include verbatim term, preferred term (PT), system organ class (SOC), treatment, severity, relationship to the interventional products, and seriousness, reporting numbers of participants experiencing each event and total numbers of each event. Laboratory safety parameters will be summarized as absolute values and changes at 28 days after each vaccination compared to baseline (before 1st vaccination) and compared to values just prior to each vaccination.

To evaluate the immunogenicity primary endpoints as defined above, SumayaVac-1 (SUM-101) vaccine induced humoral immunogenicity will be summarized as antibody responses to SumayaVac-1 (SUM-101) by ELISA over time, and fold changes of antibody responses relative to baseline.

For all analyses, data will be listed for each participant. Descriptive analyses will be performed (number of observations, arithmetic or geometric mean, standard deviation, minimum, maximum, median, interquartile range, as appropriate, for continuous data, and counts and percentages for categorical data). Results will be presented by vaccination received.

Further details will be elaborated in a Statistical Analysis Plan (SAP), including for the secondary and exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any study procedure.
2. Literate participants aged 18-45 years of African origin.
3. Female participants practicing contraception from 4 weeks before 1st immunization and both female and male participants willing to practice contraception up to 12 weeks after the last immunization.
4. Available to participate in follow-up for the duration of the study.
5. Contactable by phone during the whole study period.
6. At least two years residence in the Bagamoyo district or nearby districts in Coastal and Dar-es-Salaam regions and planning to reside there for at least 9 more months.
7. Agreement to provide personal contact information and contact information of another household member or close friend.
8. Female participants must be willing to avoid pregnancy if selected for participation in the trial and to undergo multiple serum pregnancy testing.
9. Confirmation of understanding of design, procedures, risk and benefits of the study in a test with maximum of two attempts.
10. General good health based on assessment of medical history and clinical examination.

Exclusion Criteria:

1. Previous participation in any malaria vaccine trial in the last 3 years.
2. Participation in any other clinical trial involving investigational medicinal products within 30 days prior to the screening assessment.
3. Previous history of drug or alcohol abuse interfering with normal social function within one year prior to enrolment.
4. Previous vaccination with a rabies vaccine.
5. Intake of chronic medication, especially immunosuppressive agents (steroids, immunomodulating drugs) during the 13 weeks preceding the screening visit or during the study period.
6. Known hypersensitivity to any of the vaccine components (adjuvant or protein) or anti-malarial treatments.
7. Body mass index (BMI) of <18 or >30 Kg/m2.
8. Participants unable to be closely followed for social, geographic or psychological reasons.
9. Any vaccination from 4 weeks prior to the 1st vaccination and (none planned) up to 6 weeks after the 3rd vaccination.
10. Symptoms, physical signs or laboratory values suggestive of systemic disorders, including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric and other conditions, which could interfere with the interpretation of the trial results or compromise the health of the participants.
11. Abnormal electrocardiogram on screening: pathologic Q wave and significant ST-T wave changes, left ventricular hypertrophy, clinically significant arrhythmias, left bundle branch block, secondary or tertiary A-V (atrio-ventricular) heart block.
12. Any clinically significant laboratory values at screening outside of normal ranges for study participants.
13. Malaria positivity at screening (microscopy or qPCR positive).
14. Positive HIV, HBV or HCV tests.
15. For females: Positive pregnancy test or actively breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

PRIMARY OUTCOMES:
Local and systemic adverse events (AEs) at least possibly related to the IMP after vaccination | Recorded up to 7 days after each vaccination
  Local and systemic solicited adverse events (AEs) at least possibly related to the investigational medicinal product (IMP) recorded after each vaccination (done on Day 0, Day 28 and Day 56 up to 7 days later to evaluate safety and reactogenicity of SumayaVac-1 (SUM-101)
Local and systemic unsolicited reactogenicity after vaccination | Recorded up to 28 days after each vaccination
  Local and systemic unsolicited reactogenicity recorded after each vaccination (done on Day 0, Day 28 and Day 56 up to 28 days later to evaluate the safety and reactogenicity of SumayaVac-1 (SUM-101)
Any serious adverse events (SAE) occurring after the 1st vaccination until the participant's last visit | Recorded from after 1st vaccination (Day 0 post-vaccination) until the participant's last visit (Day 140)
  Any serious adverse events (SAE) occurring after the 1st vaccination until the participant's last visit to evaluate the safety and reactogenicity of SumayaVac-1 (SUM-101)
Changes in laboratory safety parameters between baseline and 28 days after vaccination | Changes recorded between baseline (Day 0 before 1st vaccination) to 28 days after each vaccination
  Changes in laboratory safety parameters as defined in the protocol for every participant between baseline (Day 0 before 1st vaccination) to 28 days after each of the vaccinations to evaluate the safety and reactogenicity of SumayaVac-1 (SUM-101)
Changes in laboratory safety parameter prior to vaccination to 28 days after that vaccination | Changes prior to each vaccination to 28 days after proceeding with vaccination
  Changes in laboratory safety parameters as defined in the protocol for every participant between values recorded just prior to each vaccination (on Day 0, Day 28 and Day 56) and values found 28 days after proceeding with vaccination to evaluate the safety and reactogenicity of SumayaVac-1 (SUM-101)
Longevity of antibody responses to SumayaVac-1 (SUM-101) by ELISA | Titres assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit)
  Longevity of antibody responses to SumayaVac-1 (SUM-101) by ELISA for all participants at Day 0 pre-vaccination, Day 28 (Week 4), Day 56 (Week 8), Day 84 (Week 12), Day 112 (Week 16) and Day 140 (Week 20), to evaluate the humoral immunogenicity
Fold change of antibody responses to SumayaVac-1 (SUM-101) in comparison to baseline | Fold changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit)
  Fold change of antibody responses to SumayaVac-1 (SUM-101) by ELISA in comparison to baseline (Day 0 pre-vaccination) for all participants to Day 28 (Week 4), Day 56 (Week 8), Day 84 (Week 12), Day 112 (Week 16) and Day 140 (Week 20), to evaluate the humoral immunogenicity

SECONDARY OUTCOMES:
Evaluation of the opsonic phagocytosis activity of vaccine induced antibodies | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit)
  In vitro immunological assay to evaluate immune responses by measuring opsonic phagocytosis activity in the sera or blood of all participants, at Day 0 pre-vaccination, Day 28 (Week 4), Day 56 (Week 8), Day 84 (Week 12), Day 112 (Week 16) and Day 140 (Week 20).
Evaluation of complement fixation, activation and/or membrane attack complex (MAC) formation of vaccine-induced antibodies | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit)
  In vitro immunological assay to evaluate immune responses by assessing complement fixation, activation and/or membrane attack complex (MAC) formation in the sera or blood of all participants, at Day 0 pre-vaccination, Day 28 (Week 4), Day 56 (Week 8), Day 84 (Week 12), Day 112 (Week 16) and Day 140 (Week 20).
Evaluation of antibody-dependent respiratory burst (ADRB) activity of vaccine-induced antibodies | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit)
  In vitro lab immunological assay to evaluate immune responses by assessing antibody-dependent respiratory burst (ADRB) activity measured in the sera or blood of all participants, at Day 0 pre-vaccination, Day 28 (Week 4), Day 56 (Week 8), Day 84 (Week 12), Day 112 (Week 16) and Day 140 (Week 20).
Evaluation of antibody-dependent cellular cytotoxicity (ADCC-NK cells) activity of vaccine-induced antibodies | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit)
  In vitro immunological assay to evaluate immune responses by assessing antibody-dependent cellular cytotoxicity (ADCC-NK cells) activity in the sera or blood of all participants, at Day 0 pre-vaccination, Day 28 (Week 4), Day 56 (Week 8), Day 84 (Week 12), Day 112 (Week 16) and Day 140 (Week 20).
Evaluation of immune-mediated growth inhibition activity on Plasmodium falciparum asexual blood stage cell lines | Changes assessed between Day 0 (pre-vaccination) up to Day 140 (last follow up visit)
  In vitro functional assay to evaluate immune-mediated growth inhibition activity on a panel of Plasmodium falciparum asexual blood stage cell lines measured in the sera or blood of all participants, at Day 0 pre-vaccination, Day 28 (Week 4), Day 56 (Week 8), Day 84 (Week 12), Day 112 (Week 16) and Day 140 (Week 20).
Comparison of MSP-1 IgG antibody concentrations by ELISA | Antibody concentrations compared between Day 0 (pre-vaccination) up to Day 84
  Comparison of MSP-1 IgG antibody concentrations by ELISA between malaria pre-exposed participants in the current study and historical data obtained from malaria naïve participants of previous Phase Ia study conducted in Heidelberg that are assessed among SumayaVac-1 (SUM-101) participants only

OTHER OUTCOMES:
Comparison of SumayaVac-1 (SUM-101) induced immunoglobulin isotype distribution and duration | Changes observed between Day 0 (pre-vaccination) up to Day 84
  Comparison of SumayaVac-1 (SUM-101) induced immunoglobulin isotype distribution and duration in the current study and historical data obtained from malaria naïve participants of previous Phase Ia study conducted in Heidelberg that are assessed among SumayaVac-1 (SUM-101) participants only
Fine scale epitope mapping of SumayaVac-1 (SUM-101) specific antibodies | Responses measured between Day 0 (pre-vaccination) up to Day 84
  Fine scale epitope mapping of SumayaVac-1 (SUM-101) specific antibodies using peptide arrays to investigate baseline humoral responses and vaccine induced humoral responses.
Comparison of SumayaVac-1 (SUM-101) induced cellular immunity between malaria pre-exposed and malaria naïve participants from the previous Phase Ia study in Heidelberg | Changes measured between Day 0 (pre-vaccination) and Day 84
  Changes in immune cell populations between SumayaVac-1 (SUM-101) vaccinated malaria pre-exposed participants in the current trial and historical data from malaria naïve participants from the previous Phase Ia study conducted in Heidelberg including fine scale epitope mapping of MSP-1 specific CD4+ and CD8+ T cells.
Investigation of the B- and T-Cell receptor repertoire | Changes observed between Day 0 (pre-vaccination) up to Day 140
  Investigation of the B- and T-Cell receptor repertoire before and after SumayaVac-1 (SUM-101) vaccination.
Cellular immune responses to SumayaVac-1 (SUM-101) | Changes observed between Day 0 (pre-vaccination) and Day 56 (W8), Day 84 (W12), Day 112 (W16) and Day 140 (W20).
  Cellular immune responses to SumayaVac-1 (SUM-101) by (i) ELISpot assays using total PBMC, (ii) SumayaVac-1 (SUM-101) specific cells characterised by flow cytometry-based immunophenotyping using intracellular cytokine staining (ICS), (iii) functional gene expression analysis, and/or other assays to be defined; at D0 pre-vac and D56 (W8), D84 (W12), D112 (W16) and D140 (W20).
Integrated transcriptome and immunoglobulin gene repertoire analyses | Changes observed between Day 0 (pre-vaccination) up to Day 140
  Integrated transcriptome and immunoglobulin gene repertoire analyses of MSP-1 specific B-cells using single-cell technologies before and after SumayaVac-1 (SUM-101) vaccination.
Glycosylation patterns of MSP-1 specific functional antibodies | Changes observed between Day 0 (pre-vaccination) up to Day 84
  Lab based assays to assess the glycosylation patterns of MSP-1 specific functional antibodies.
Investigate off-target IgG and IgM repertoire after SumayaVac-1 (SUM-101) vaccination | Changes observed between Day 0 (pre-vaccination) up to Day 140
  Investigate off-target IgG and IgM repertoire after SumayaVac-1 (SUM-101) vaccination using immunoproteomics.
Investigate the structure of recombinant MSP-1 protein bound to functional antibodies | Through study completion, an average of 1 year
  Investigate the structure of MSP-1 protein bound to functional antibodies by cryo-electron tomography to map conformational epitopes
Ex vivo assessment of changes in human peripheral blood transcriptome | Changes observed between Day 0 (pre-vaccination) and Day 140
  Ex vivo assessment of changes in human peripheral blood transcriptome in participants having received SumayaVac-1 (SUM-101) versus Verorab® rabies vaccine.
Description of ɣδ T-cell receptor repertoire, transcriptome, functional activity and phenotypes | Changes observed between Day 0 (pre-vaccination) and Day 140
  Description of ɣδ T-cell receptor repertoire, transcriptome, functional activity and phenotypes in participants having received SumayaVac-1 (SUM-101) versus Verorab® rabies vaccine.
Investigate the impact of the presence of intestinal helminth infections on vaccine-induced humoral immune response | Changes observed between Day 0 (pre-vaccination) and Day 84
  Investigate the impact of the presence of intestinal helminth infections on vaccine-induced humoral immune response by comparing the quality and quantity of SumayaVac-1 (SUM-101) specific antibody isotypes between helminth infected and non-infected participants at baseline
Investigate the impact of the presence of intestinal helminth infections on SumayaVac-1 (SUM-101) vaccine-induced cellular immune responses | Changes observed between Day 0 (pre-vaccination) and Day 84
  Investigate the impact of the presence of intestinal helminth infections on SumayaVac-1 (SUM-101) vaccine-induced cellular immune responses by comparing the quality and quantity of SumayaVac-1 (SUM-101) specific cytokine production and ICS results between helminth infected and non-infected participants at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Daubenberger, PhD, Study Chair — Swiss Tropical & Public Health Institute; Ally Olotu, MD, Principal Investigator — Ifakara Health Institute
Locations (1):
- Ifakara Health Institute, Bagamoyo, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blank A, Furle K, Jaschke A, Mikus G, Lehmann M, Husing J, Heiss K, Giese T, Carter D, Bohnlein E, Lanzer M, Haefeli WE, Bujard H. Immunization with full-length Plasmodium falciparum merozoite surface protein 1 is safe and elicits functional cytophilic antibodies in a randomized first-in-human trial. NPJ Vaccines. 2020 Jan 31;5(1):10. doi: 10.1038/s41541-020-0160-2. eCollection 2020. PMID 32025341
- [Derived] Kahatano AE, Mpina M, Vanobberghen F, Hassan O, Urasa N, Sasamalo I, Mswata S, Paris D, Gajewski S, Saxena M, Furle K, Kiehl V, Bohnlein E, Aschenbrenner A, Lanzer M, Thomson-Luque R, Olotu A, Daubenberger C. Full-length merozoite surface protein 1 formulated with GLA-SE adjuvant in malaria pre-exposed adults: a randomised, controlled, double-blind, parallel-group, single-centre Phase Ib trial. EClinicalMedicine. 2025 Oct 25;89:103585. doi: 10.1016/j.eclinm.2025.103585. eCollection 2025 Nov. PMID 41210385
- See also: Related Info — https://www.nature.com/articles/s41541-020-0160-2